CLINICAL TRIAL: NCT02171130
Title: A Multiple Center, Open Label, Prospective, Observational Study to Evaluate the Effectiveness and Ease-of-Use of AMG504-1 Administered in the Home or Work Environments for Treating Episodes of Hypoglycemia in Patients With Type 1 Diabetes
Brief Title: Clinical Usability of Intranasal Glucagon in Treatment of Hypoglycemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Locemia Solutions ULC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16427; I8R-MC-B002 (Other: Eli Lilly and Company); AMG108 (Other: Locemia Solutions ULC)
Record Dates: First submitted 2014-06-12; First posted 2014-06-24 (Estimated); Results first posted 2019-10-15 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2017-03

CONDITIONS: Hypoglycemia; Diabetes Mellitus; Drug-Specific Antibodies
Keywords: Diabetes Mellitus; Hypoglycemia; Glucagon; Anti-glucagon Antibody; Immunogenicity
MeSH Terms: conditions — Hypoglycemia; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nasal glucagon (Experimental): 3 mg nasal glucagon powder delivered using a nasal powder dosing device.
  Interventions: Drug: Nasal Glucagon

INTERVENTIONS:
Drug: Nasal Glucagon — 3 mg nasal glucagon powder
  Other Names: Dry-Mist Nasal Glucagon; AMG504-1; LY900018

SUMMARY:
Up to two hundred (200) adult participants with type 1 diabetes (T1D) aged 18 to 75 years will be selected for inclusion in the study. The target is to obtain treatment response and user-experience data following use of nasal glucagon (AMG504-1) in treating episodes of hypoglycemia. The population will be enriched to include participants who suffer from impaired hypoglycemia awareness.

DETAILED DESCRIPTION:
This study is designed to evaluate the effectiveness of nasal glucagon (NG) administered under clinical use conditions in treating episodes of hypoglycemia in persons with T1D.

This study also aims to assess the ease with which caregivers can administer the experimental medication in treatment of hypoglycemic events.

The study will also generate data on the participants' assessment of local tolerability and provide information on immunogenicity of nasal glucagon with regards to the potential development of anti-glucagon antibodies.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female Person with diabetes (PWD) lives with or is in frequent contact with one or more caregivers who are available to administer the glucagon in case of an episode of severe or moderate hypoglycemia
* With a history of type 1 diabetes >1 year
* At least 18 years of age but not older than 75 years
* Body mass index (BMI) greater than or equal to 18.50 and below 35.00 kg/m2.
* PWD will be otherwise healthy according to medical history, general physical examination (including vital signs), nasal examination, and laboratory tests (biochemistry, hematology, and urinalysis).
* For female subjects, a urine pregnancy test must be negative.

Exclusion Criteria:

* Presence or history of pheochromocytoma (i.e. adrenal gland tumor) or insulinoma.
* Use of a daily systemic beta-blockers, indomethacin, warfarin or anticholinergic drugs.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2014-05; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (9):
- United States (3):
  - New England Diabetes and Endocrinology Center (NEDEC), Waltham, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Albany Medical College Division of Community Endocrinology, Albany, New York
- Canada (6):
  - Winnipeg Clinic, Winnipeg, Manitoba
  - Diabetes Clinic, Smiths Falls, Ontario
  - IRCM, Montreal, Quebec
  - Centre Hospitalier de l'Université de Québec, Québec, Quebec
  - Centre de recherche d'endocrinologie Godin & St-Pierre, Sherbrooke, Quebec
  - Applied Medical Informatics Research, Westmount, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants and their principal caregiver(s) were trained in the use of nasal glucagon.
Groups:
- Nasal Glucagon (NG): Nasal Glucagon powder (3 milligram [mg])
Period: Overall Study
Arm/Group | Nasal Glucagon (NG)
Started | 129
Received at Least One Dose of Study Drug | 87
Experienced Hypoglycemic Event | 87 (Experienced at least one hypoglycemic event and received at least one dose of study drug.)
Completed | 101 (Including participants who completed the 6-month study but did not experience any hypoglycemia event)
Not Completed | 28
Not completed — Death | 1
Not completed — Discontinued; Clinical Material Issue | 16
Not completed — Discontinued; Site Termination | 5
Not completed — Withdrawal by Subject | 3
Not completed — Physician Decision | 1
Not completed — Lost to Follow-up | 1
Not completed — Met Exclusion Criteria | 1

BASELINE CHARACTERISTICS:
Groups:
- Nasal Glucagon: Nasal Glucagon powder (3mg)
Arm/Group | Nasal Glucagon
Number analyzed (Participants) | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.6 (14.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56
  Male | 73
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 123
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 81
  United States | 48

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Awakening or Returning to a Normal Status Within 30 Minutes Following Studied Drug of Administration
Description: Responses to questions completed by the caregiver were used to assess this outcome.
  An episode of severe hypoglycemia was defined as an episode wherein the person with diabetes is clinically incapacitated to the point where the person requires third-party assistance to treat the hypoglycemia. An episode of moderate hypoglycemia episode was defined as an episode wherein the person with diabetes was showing signs of neuroglycopenia and had a glucometer reading of approximately 60 milligrams per deciliter (mg/dL) (3.3 millimoles per liter [mmol/L]) or less based on a blood sample taken at or near the time of treatment.
Time Frame: Within 30 minutes after each drug administration for an episode of hypoglycemia
Population: Enrolled participants received at least 1 dose of the study drug with evaluable hypoglycemic event. Events requiring additional medical assistance or rescue therapy within 30 minutes of study drug administration and participants from a Good Clinical Practice (GCP) non-compliant site were excluded.
Measure: Number; unit: percentage of participants
Arm/Group | Nasal Glucagon
Number analyzed (Participants) | 69
percentage of participants | 95.7

2. Secondary Outcome: Assessment of Ease-of-use of Dry-Mist Nasal Glucagon as Determined by Completion of Questionnaires by the Caregiver
Description: Measurement for Degree of difficulty: opening the kit, Degree of difficulty: understanding the instructions on how to use the kit, Degree of difficulty: administering the medication into the nostril, Degree of satisfaction is 1 (Very Difficult) to 7 (Very Easy). Measurement for Dry Mist Nasal Glucagon will be easy to teach other caregivers, Nasal formulation of glucagon is less intimidating for caregivers, Nasal Glucagon is easy to carry and would be willing to carry it, nasal delivery of glucagon is preferable. Level of agreement 1 (Strongly Disagree) to 7 (Strongly Agree).
Time Frame: After each drug administration for an episode of hypoglycemia
Population: Eligible enrolled participants who experienced at least 1 hypoglycemic event and received at least 1 dose of study drug. Participants from the GCP non-compliant site and participants who were impacted by a clinical material issue which might have led to under-dose, were considered ineligible thus excluded from this population.
Measure: Count of Units; unit: Total Number of Events
Units Other Than Participants: Total Number of Events
Arm/Group | Nasal Glucagon
Number analyzed (Participants) | 74
Number analyzed (Total Number of Events) | 179
Total Number of Events
  Difficulty: opening the kit (Very Difficult) | 2
  Difficulty: opening the kit (Average) | 4
  Difficulty: opening the kit (Relatively Easy) | 4
  Difficulty: opening the kit (Easy) | 26
  Difficulty: opening the kit (Very Easy) | 143
  Difficulty: instructions (Very Difficult) | 2
  Difficulty: instructions (Average) | 4
  Difficulty: instructions (Relatively Easy) | 10
  Difficulty: instructions (Easy) | 36
  Difficulty: instructions (Very Easy) | 127
  Difficulty: administering (Very Difficult) | 4
  Difficulty: administering (Relatively Difficult) | 7
  Difficulty: administering (Average) | 8
  Difficulty: administering (Relatively Easy) | 16
  Difficulty: administering (Easy) | 42
  Difficulty: administering (Very Easy) | 102
  Time to administer (<30 seconds) | 126
  Time to administer (30-<60 seconds) | 40
  Time to administer (1-<2 minutes) | 9
  Time to administer (2-<5 minutes) | 4
  Degree of satisfaction (Relatively Difficult) | 3
  Degree of satisfaction (Average) | 7
  Degree of satisfaction (Relatively Easy) | 21
  Degree of satisfaction (Easy) | 48
  Degree of satisfaction (Very Easy) | 100
  Compare to Injectable (Not Applicable) | 108
  Compare to Injectable (Much Easier) | 47
  Compare to Injectable (Easier) | 4
  Compare to Injectable (Missing) | 20
  Ease to teach other (Neither Agree nor Disagree) | 2
  Ease to teach other (Somewhat Agree) | 3
  Ease to teach other (Mostly Agree) | 47
  Ease to teach other (Strongly Agree) | 127

3. Secondary Outcome: Percentage of Participants With Adverse Events (AEs) Reported Through the Nasal Score Questionnaire
Description: Adverse events solicited through the Nasal Score Questionnaire included: runny nose, nasal congestion (nostrils plugged), nasal itching, sneezing, watery eyes, itchy eyes, redness of eyes, itching of ears, itching of throat, and other.
  A summary of other nonserious AEs, and all Serious Adverse Events (SAEs), regardless of causality, is located in the Reported Adverse Events section.
Time Frame: Within 2 hours of full recovery from a hypoglycemic event
Population: Eligible enrolled participants who experienced at least 1 hypoglycemic event and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Nasal Glucagon
Number analyzed (Participants) | 87
percentage of participants | 82.8

4. Other Pre Specified Outcome: Blood Glucose Levels Over Time
Description: The participants' blood glucose level was measured by the caregiver using a glucometer at baseline (just prior to dosing and right after the study drug administration), 15, 30 and 45 minutes after nasal glucagon administration.
Time Frame: Baseline (just prior to dosing or right after study drug administration) , 15, 30 and 45 minutes after drug administration for an episode of hypoglycemia
Population: Enrolled participants received at least 1 dose of the study drug with evaluable hypoglycemic event. Events requiring additional medical assistance or rescue therapy within 30 minutes of study drug administration and participants from a GCP non-compliant site were excluded.
Measure: Mean (Standard Deviation); unit: milligram/deciliter (mg/dL)
Units Other Than Participants: Total Number of Hypoglycemic Events
Arm/Group | Nasal Glucagon
Number analyzed (Participants) | 69
Number analyzed (Total Number of Hypoglycemic Events) | 157
milligram/deciliter (mg/dL)
  Baseline | 47.9 (10.47)
  15 minutes drug administration | 84.4 (24.68)
  30 minutes drug administration | 112.8 (34.33)
  45 minutes drug administration | 123.1 (38.82)

5. Other Pre Specified Outcome: Number of Participants With Treatment-Emergent Glucagon Anti-Drug Antibodies (ADA)
Description: Treatment-Emergent ADA includes treatment-induced ADA ('Not Detected' ADA at baseline and at least one post-baseline 'Detected' ADA sample with a corresponding titer of (1:20) and treatment-boosted ADA (with 'Detected' ADA at baseline and at least one post-baseline 'Detected' ADA sample with a corresponding titer that is at least 4-fold higher than the baseline titer.
Time Frame: Baseline and End of Study (6 months)
Population: Enrolled participants who had antibody sample at both baseline and post-baseline.
Measure: Number; unit: percentage of participants
Arm/Group | Nasal Glucagon
Number analyzed (Participants) | 43
percentage of participants | 0

ADVERSE EVENTS:
Time Frame: After study drug administration, up to 6 months.
Description: Adverse events were collected systematically using the Hypoglycemia Questionnaire.
  Analysis population included participants with at least one exposure to study drug after hypoglycemic event.
Arm/Group | Nasal Glucagon
All-Cause Mortality (participants affected / at risk) | 1/87
Serious Adverse Events (participants affected / at risk) | 1/87
Other Adverse Events (participants affected / at risk) | 74/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nasal Glucagon (N=87)
Death (General disorders) | 1 (1) — This death was due to Klebsiella pneumoniae infection and not related to study drug.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nasal Glucagon (N=87)
Ear pain (Ear and labyrinth disorders) | 5 (6)
Eye inflammation (Eye disorders) | 1 (1)
Eye pain (Eye disorders) | 2 (3)
Hypoaesthesia eye (Eye disorders) | 1 (1)
Lacrimation increased (Eye disorders) | 8 (10)
Asthenia (General disorders) | 1 (1)
Facial pain (General disorders) | 1 (1)
Feeling abnormal (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Product taste abnormal (General disorders) | 3 (3)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Burning sensation (Nervous system disorders) | 1 (1)
Head discomfort (Nervous system disorders) | 1 (1)
Sinus headache (Nervous system disorders) | 2 (2)
Somnolence (Nervous system disorders) | 1 (2)
Choking (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 20 (29) — Hypoglycemia Questionnaire
Vomiting (Gastrointestinal disorders) | 8 (16) — Hypoglycemia Questionnaire
Nasal Irritation (Respiratory, thoracic and mediastinal disorders) | 67 (117) — Hypoglycemia Questionnaire
Headache (Nervous system disorders) | 45 (72) — Hypoglycemia Questionnaire

LIMITATIONS AND CAVEATS:
Sixteen participants were discontinued early because of a clinical trial material issue which might have led to under-dose. One site was terminated due to GCP non-compliance and five participants were discontinued as a result.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days